CLINICAL TRIAL: NCT00892372
Title: Relationship Between Changes in Body Weight and Glycohemoglobin Levels in Patients With Type 2 Diabetes Treated With Diet or Pioglitazone.
Brief Title: Relationship Between Body Weight and Glycohemoglobin
Status: Completed | Type: Observational
Sponsor: Saitama Medical University (Other)
Responsible Party: Eiji Ohmura/ M.D., Saitama Medical center, Saitama Medical University
Other Study IDs: bwhba1c
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: body weight; glycohemoglobin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body Weight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 (type 2 diabetes, body weight, HbA1c): The investigators analyzed the recorded data (body weight and glycohemoglobin) of 70 type 2 diabetic patients treated with the diet therapy. Recorded values at 0, 2 and 4 months for body weight (BW) and glycohemoglobin (HbA1c) were used. And changes from baseline (0 month) in BW (ΔBW) were plotted against those of HbA1c (ΔHbA1c).
- 2 (type 2 diabetes, pioglitazone, HbA1c): The investigators analyzed the recorded data (body weight and glycohemoglobin) of 23 type 2 diabetic patients treated with pioglitazone. Recorded values at 0, 2 and 4 months for body weight (BW)and glycohemoglobin (HbA1c) were used. And changes from baseline (0 month) in BW (ΔBW) were plotted against those of HbA1c (ΔHbA1c).

SUMMARY:
Control of body weight (BW) is important to prevent and manage type 2 diabetes. Regardless of the close association, little is understood about the precise relationship between BW and glycemic control, which might be of benefit for patients with type 2 diabetes. The researchers investigated the correlation between changes in BW and glycemic control in patients with type 2 diabetes treated with a diet therapy or pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes under reasonable glycemic control (HbA1c; less than around 7%)
* type 2 diabetic patients treated with the diet therapy

Exclusion Criteria:

* type 2 diabetic patients with edema, severe liver dysfunction, renal dysfunction, moderate to severe anemia or congestive heart failure
* type 2 diabetic patients treated with insulin therapy

Ages: 32 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Ohmura, M.D., Principal Investigator — Department of Diabetes and Endocrinology, Saitama Medical Center, Saitama Medical University
Locations (1):
- Department of Diabetes and Endocrinology, Saitama Medical Center, Saitama Medical University, Kawagoe, Saitama, Japan